CLINICAL TRIAL: NCT01818167
Title: A Prospective Multi-Center Blinded, Randomized, Controlled Clinical Trial Comparing the Efficacy of Provodine Topical Body Wash Versus 10% Benzoyl Peroxide Topical Body Wash for the Treatment of Hidradenitis Suppurativa
Brief Title: An Investigation Into the Efficacy of Provodine Topical Cream as Compared to 10% Benzoyl Peroxide Wash for the Treatment of Hidradenitis Suppurativa.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Microdermis Corporation (Industry)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Microdermis-100
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; HS; Acne Inversa; Velpeau's disease; Verneuil's disease
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% Benzoyl Peroxide Topical Body Wash (Active Comparator): Subjects will use 10% benzoyl peroxide twice daily. The product will be applied to the affected areas, left on for 45 seconds, then rinsed off.
  Interventions: Drug: 10% Benzoyl Peroxide Topical Body Wash
- Provodine Topical Cream (Active Comparator): Subjects will use Provodine Topical Cream twice daily. The product will be applied to the affected areas, left on for 45 seconds, then rinsed off.
  Interventions: Drug: Provodine Topical Cream

INTERVENTIONS:
Drug: 10% Benzoyl Peroxide Topical Body Wash
  Arms: 10% Benzoyl Peroxide Topical Body Wash
Drug: Provodine Topical Cream
  Arms: Provodine Topical Cream

SUMMARY:
The purpose of this study is to compare the efficacy of Provodine™ topical cream to 10% benzoyl peroxide topical body wash for the treatment of early stage hidradenitis suppurativa.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, recurrent inflammatory disease of the skin. It typically manifests as nodules and abscesses that ultimately can progress to form deep sinus tracts, fistulas, and scarring. It affects areas of the body with apocrine gland bearing tissue, including the anogenital, axillary and inframammary regions. The lesions are often very painful and can chronically drain malodorous fluid, which can leave affected individuals uncomfortable and self-conscious, or even debilitated. The pathogenesis of this disease process is not fully understood, and the HS can be difficult to treat. Measures such as topical antibiotic and antiseptic washes are generally thought to be beneficial for the treatment of early stage HS. Although there have been no controlled trials for the treatment of HS, commonly used topical washes currently include benzoyl peroxide and chlorhexidine gluconate.

Provodine™ topical cream was designed to actively kill microbes on the skin for up to 6 hours without resulting in the irritation often associated with repetitive use of antimicrobial products. A blinded controlled comparison of Provodine™ versus the current standard of benzoyl peroxide wash will not only allow for an alternative treatment for early stage HS but also provide an additional tool in the arsenal of treatments for this disease process.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion, the subject must:

  1. Be at least 13 years old.
  2. Be otherwise healthy.
  3. Have a diagnosis of HS.
  4. Patients must have Hurley stage I or Stage II HS
  5. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form.
  6. Agree to follow and undergo all study-related procedures.
  7. If applicable, minors must have permission of legal guardian for participation in the study.

Exclusion Criteria:

* Subjects who meet the following criteria will be excluded:

  1. Patients with HS Hurley stage III will be excluded from participation in the study
  2. Patients who are pregnant or breast feeding will not be able to take part in the study due to the unknown effects of the topical medications.
  3. Concomitant use of systemic or other topical treatments for HS not involved in current study. For cohort I, no washout period for systemic and/or topical medications will be required. For Cohort II, there will be a 14 day minimum washout period for systemic and topical treatments for HS.
  4. Any reason the investigator feels the patient should not participate in the study.
  5. If a patient misses ≥ 2 consecutive study visits, the patient will be excluded from further participation in this trial.
  6. History of allergy to iodine or benzoyl peroxide.

Ages: 13 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01-05 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-01-21 (Actual)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa European Research Group (HISERG) scale | 4 months
  Assessment of the degree of involvement of HS will be performed at each study visit using the Hidradenitis Suppurativa European Research Group (HISERG) scale outlined below:
  1. Anatomical region involved (axilla, groin, gluteal or other region or inframammary region left and/or right: 3 points per region involved).
  2. Number and scores of lesions (abscesses, nodules, fistulas, scars: points per lesion of all regions involved: nodules 2, fistulas 4, scars 1, others 1)
  3. The longest distance between two relevant lesions, i.e., nodules and fistulas, in each region, or size if only one lesion (<5cm 2, <10cm 4, >10cm 8)
  4. Are all lesions clearly separated by normal skin? In each region (yes 0/no 6)
  5. Extent of erythema, edema, pain and purulent discharge of each anatomic site (0-3 for each clinical indicator)

SECONDARY OUTCOMES:
Skin Irritation Index | 4 months
  Subjects will be evaluated weekly for any signs or symptoms of local skin irritation by a study physician using the following Skin Irritation Index scoring system, which includes ratings for erythema, edema, scaling and dryness, rash and discomfort.
Patient reported Quality of Life Scores on the Dermatology Quality of Life Index and the Skindex-20 | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Dermatology
Locations (1):
- Henry Ford Medical Center Department of Dermatology, Detroit, Michigan, United States